CLINICAL TRIAL: NCT04626440
Title: Comprehensive Precision Medicine Research on the Heterogeneity of Taiwanese Breast Cancer Patients by Next Generation Sequencing (NGS) Tools
Brief Title: Research on the Heterogeneity of Taiwanese Breast Cancer Patients by Next Generation Sequencing (NGS) Tools
Status: Recruiting | Type: Observational
Sponsor: vghtpe user (Other Government)
Collaborators: YongLin Healthcare Foundation (Unknown)
Responsible Party: Sponsor-Investigator, vghtpe user, Chief of Comprehensive Breast Health Center, Department of Surgery, Taipei Veterans General Hospital, Taiwan
Organization: Taipei Veterans General Hospital, Taiwan (Other Government)
Other Study IDs: 2018-09-007A; QCR18002 (Other Grant/Funding Number: YongLin Healthcare Foundation)
Record Dates: First submitted 2020-11-02; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Next Generation Sequencing (NGS); Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Group 1 [(A) subjects who are planning to receive surgery (mastectomy or BCS) as the first-line treatment for BC and followed by adjuvant therapy, or (B) subjects with BC recurrence at screening, who had received surgery for primary BC within 3 years prior to screening, and with primary tumor FFPE tissues available]
  Interventions: Procedure: Diagnostic stage or the Clinical outcome
- Group 2: subjects who are planning to receive neoadjuvant therapy as the first-line treatment for BC and followed by surgery
  Interventions: Procedure: Diagnostic stage or the Clinical outcome
- Group 3: Group 3-1 (subjects diagnosed with de novo and treatment naïve stage IV BC); or Group 3-2 [(A) stage IV subjects with BC recurrence beyond 3 years after surgery (mastectomy or BCS) or stage IV subjects who had received or are currently receiving treatments for BC].
  Interventions: Procedure: Diagnostic stage or the Clinical outcome

INTERVENTIONS:
Procedure: Diagnostic stage or the Clinical outcome — After enrollment, individual subject will be assigned into one of the four groups according to the medical management received, the diagnostic stage of breast cancer (BC), or the clinical outcome of BC at enrollment.

SUMMARY:
The objectives of this study are:

1. To determine the difference in genetic profiling of subjects with breast cancer recurrence
2. To determine the comprehensive genetic profiling of subjects with late stage breast cancer
3. To determine the potential biomarkers for early detection and prognosis for breast cancer
4. To determine the genetic profiling of immune system in different subtypes of breast cancer

By integrating and analyzing the data generated using the methods of NGS, these information can be used for:

1. Understanding the genetic profiling of different subtypes of breast cancer in Taiwan
2. Assessing the efficacy of different treatments in breast cancer subjects
3. Defining the molecular risk factors and predicting the potential risk of breast cancer recurrence
4. Assessing the immune repertoire and the potential effects of immunotherapy in breast cancer subjects
5. Developing new strategies in treating patients with triple negative or late stage of breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged over 20 years old
* Subject with confirmed diagnosis of primary invasive breast cancer and is planning to receive treatments for breast cancer. However, subjects with breast cancer recurrence at screening will be enrolled if meet both the following conditions:

  1. Subjects had received surgery for primary breast cancer within 3 years prior to screening [i.e. recurrence within 3 years after surgery (mastectomy or BCS)];
  2. Subjects diagnosed with stage IV breast cancer beyond 3 years after surgery (mastectomy or BCS) or who had received or are currently receiving treatments for breast cancer. And subjects with primary tumor FFPE tissues available and pass the RNA quality check.
* Eastern Cooperative Oncology Group (ECOG) Performance score ≤ 3
* Life expectancy ≥ 3 months
* Subject agrees to provide the written informed consent. If a subject has breast cancer recurrence within 3 years prior to screening, she will be eligible if she agrees to provide the paired FFPE tissues (primary and recurrent tumors)

Exclusion Criteria:

* Subjects will be excluded if they had primary cancer other than breast cancer within 5 years prior to screening

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with confirmed diagnosis of primary invasive breast cancer and is planning to receive treatments for breast cancer.
Sampling Method: Probability Sample
Enrollment: 1875 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The rate of genomic alteration | Aug.2026
  Discovery of comprehensive genetic profiles including copy number variation and single nucleotide polymorphism in group 1, 2 and 3 subjects.
  Discovery of genetic mutations of T cell receptor
Clinical outcome | Aug.2026
  Breast cancer recurrence, overall survival and recurrence-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu CY, Huang CC, Tsai YF, Chao TC, Lien PJ, Lin YS, Feng CJ, Chen JL, Chen YJ, Chiu JH, Hsu CY, Tseng LM. VGH-TAYLOR: Comprehensive precision medicine study protocol on the heterogeneity of Taiwanese breast cancer patients. Future Oncol. 2021 Oct 19. doi: 10.2217/fon-2021-0131. Online ahead of print. PMID 34665002